CLINICAL TRIAL: NCT04755530
Title: Matrix Characterization and Effects of Fermented Dairy Products on Liver Fat, Cardiometabolic Risk and Gut Microbiome in Males With Symptoms of Metabolic Syndrome
Brief Title: Fermented Dairy Products and The Metabolic Syndrome
Acronym: FerMetS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faidon Magkos (Other)
Collaborators: Arla Food for Health (Unknown); University of Aarhus (Other); Mælkeafgiftsfonden (Unknown); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Faidon Magkos, Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B363; H-20059243 (Registry Identifier: Danish Ethical Committee)
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Overweight or Obesity; Metabolic Syndrome
Keywords: Dairy; Liver fat; Glucose metabolism
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome; Fatty Liver | interventions — Dairy Products; Milk; Yogurt; Cultured Milk Products

STUDY DESIGN:
Intervention Model Description: 16-week parallel randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Until the statistical analyses are performed, principal investigator and statistician are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Regular whole milk (Active Comparator): Substitution of a part of the habitual diet with 400 g/day of regular whole milk
  Interventions: Dietary Supplement: Regular whole milk
- Yogurt with live bacteria (Experimental): Substitution of a part of the habitual diet with 400 g/day of yogurt with life bacteria
  Interventions: Dietary Supplement: Yogurt with live bacteria
- Yogurt with inactivated bacteria (Experimental): Substitution of a part of the habitual diet with 400 g/day of yogurt with inactivated bacteria
  Interventions: Dietary Supplement: Yogurt with inactivated bacteria
- Acidified whole milk (Experimental): Substitution of a part of the habitual diet with 400 g/day of acidified whole milk
  Interventions: Dietary Supplement: Acidified whole milk

INTERVENTIONS:
Dietary Supplement: Regular whole milk — 400 g/day of regular whole milk
  Other Names: Dairy product; Milk
  Arms: Regular whole milk
Dietary Supplement: Yogurt with live bacteria — 400 g/day of yogurt with live bacteria
  Other Names: Fermented dairy product; Yogurt
  Arms: Yogurt with live bacteria
Dietary Supplement: Yogurt with inactivated bacteria — 400 g/day of yogurt with inactivated bacteria
  Other Names: Fermented dairy product; Yogurt
  Arms: Yogurt with inactivated bacteria
Dietary Supplement: Acidified whole milk — 400 g/day of yogurt with acidified whole milk
  Other Names: Dairy product
  Arms: Acidified whole milk

SUMMARY:
The study will be conducted as a randomized controlled trial with four parallel arms including four dairy products. We will investigate the health effects of including yogurt in the diet through a 16-weeks intervention period among 100 volunteering males with symptoms of the metabolic syndrome. The study has a total duration of 20 weeks as a wash out period of four weeks will be initiated prior to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Age between 30-70 years
* BMI of 28-45 kg/m2
* Abdominal obesity (defined as waist circumference >102 cm)
* Provided voluntary written informed consent

Exclusion Criteria:

* Body weight changes +/- 5% in the past three months
* Any diet, allergy or intolerance which results in not being able to follow the study protocol
* Contraindications related to MRI (pacemaker, stent, magnitic metal in the body, claustrophobia, physiological diseases or a body weight >160 kg)
* History or diagnosis of diabetes
* History or diagnosis of heart, liver, gastrointestinal or kidney disease
* History or diagnosis of illness related to energy balance
* History or diagnosis of eating disorders
* Simultaneous blood donation for other purpose than this study (and one month before initiating the study)
* Simultaneous participation in other clinical intervention studies
* Any other condition that judged by the investgator may interfere with the adherence to the study protocol

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on self-representation of gender identity
Enrollment: 100 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Liver fat | Change from Week 0 to week 16
  Measurements of liver fat by Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Cardiometabolic risk | Change from Week 0 to week 16
  Measured by fasting cholesterol, HDL, LDL, Triglycerid and LDL fractions
Cardiometabolic risk | Change from Week 0 to week 16
  Measured by fasting ALAT
Cardiometabolic risk | Change from Week 0 to week 16
  Measured by fasting blood pressure (automatic device)
Gut microbiome | Change from week -4 to week 16
  Measurments of microbiota (fecal spot samples)
Glucose metabolism (fasting samples) | Change from Week 0 to week 16
  Measurements of fasting glucose, insulin, C-peptide, HbA1C
Glucose metabolism (5 hour oral glucose tolerance test) | Week 16 (5 hour test)
  Measurements of glucose, insulin and C-peptide during a 5 hour oral glucose tolerance test
Inflammation | Change from Week 0 to week 16
  Measurements of fasting CRP
Inflammation | Change from Week 0 to week 16
  Measurements of fasting IL-6
Inflammation | Change from Week 0 to week 16
  Measurements of fasting TNF-alfa
Body composition | Change from week -4 to week 16
  Measurements of body weight (every week), height (stadiometer) (only at screening), waist and hip circumference (non-elastic tape), sagittal diameter (abdominal caliper) (only week 0 and 16) as wells as fat mass and fat free mass (whole body DXA scan) (only week 0 and 16).
Fat disposition and pancreatic fat | Change from Week 0 to week 16
  Measurements of viceral, subcutaneous and pancreatic fat by Magnetic Resonance Imaging

OTHER OUTCOMES:
Metabolome | Change from week -4 to week 16
  Measurement of metabolomic markers in blood, urine and feces
Physical activity | Change from week -4 to week 16
  Measured by International Physical Activity Questionnaire (IPAQ)
Sleep quality | Change from week -4 to week 16
  Measured by Pittsburg Sleep Quality Index (PSQI)
Perceived stress | Change from week -4 to week 16
  Measured by Perceived Stress Scale (PSS)
Life quality | Change from week -4 to week 16
  Measured by Physical and mental life quality, Short Form-36 (SF-36)
The influence of initial glucose metabolism | Change from week -4 to week 16
  Statistical investigation of the effect of initial glucose metabolism on liver fat
The influence of initial gut microbiota | Change from week -4 to week 16
  Statistical investigation of the effect of initial microbiota assessed by fecal sample on liver fat
The influence of initial body composition | Change from week -4 to week 16
  Statistical investigation of the effect of initial body composition assessed by DXA scan on liver fat

CONTACTS AND LOCATIONS:
Overall Officials: Faidon Magkos, PhD, Principal Investigator — University of Copenhagen, Department of Nutrition, Exercise and Sports
Locations (1):
- University of Copenhagen, Department of Nutrition, Exercise and Sports, Frederiksberg, DK, Denmark

REFERENCES:
- [Derived] Sandby K, Magkos F, Chabanova E, Petersen ET, Krarup T, Bertram HC, Kristiansen K, Geiker NRW. The effect of dairy products on liver fat and metabolic risk markers in males with abdominal obesity - a four-arm randomized controlled trial. Clin Nutr. 2024 Feb;43(2):534-542. doi: 10.1016/j.clnu.2023.12.018. Epub 2023 Dec 27. PMID 38232682